CLINICAL TRIAL: NCT05890807
Title: Evaluation of the Concordance in the Diagnosis of Periodontitis in Diabetic Patients Between an Indirect Method Based on a Photograph of the Oral Cavity and a Direct Method Based on the Clinical Examination of This Oral Cavity (Reference).
Brief Title: Concordance in Diagnosis of Periodontitis in Diabetic Patients Between an Indirect Method Based on a Photograph of the Oral Cavity and a Direct Method Based on the Clinical Examination of This Oral Cavity (Reference).
Acronym: PARODIABNOSTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A02129-34
Record Dates: First submitted 2023-05-15; First posted 2023-06-06 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Complications; Periodontal Diseases
Keywords: Diabetes; Periodontitis
MeSH Terms: conditions — Diabetes Complications; Periodontal Diseases; Diabetes Mellitus; Periodontitis

STUDY DESIGN:
Intervention Model Description: A prospective, single-center, open-label, cross-sectional study to evaluate the concordance of an intervention versus the "gold standard.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients whose oral cavity will be photographed in the diabetology department (Experimental): The patient is seated in the chair. The trained staff member positions the mouth guard and takes a frontal photograph of the patient's oral cavity using the photo sensor (smart-phone). Only the oral cavity will be visible in the photograph and there will be no possibility for an external assessor to recognize the patient's face.
  Interventions: Diagnostic Test: Front view photography of the patient's oral cavity with the help of a smartphone in the diabetology department.

INTERVENTIONS:
Diagnostic Test: Front view photography of the patient's oral cavity with the help of a smartphone in the diabetology department. — The diabetologist will take a photograph of the patient's oral cavity in the diabetology department.

SUMMARY:
Periodontitis, a known complication of diabetes, is an infectious disease that destroys bone and gums. Studies have shown that diabetes favors periodontitis, and that periodontitis contributes to its aggravation. The positive impact of treating periodontitis on the cost of diabetes care has been demonstrated and the French national health system fully covers the treatment of periodontitis for diabetic patients. Unfortunately, 80% of diabetic patients do not visit their dentist enough.

Although diabetologists regularly see their patients and are aware of the importance of treating periodontitis,they do not have the expertise to diagnose the condition whereas a specialist dentist can often diagnose it just by looking.

This study aims to develop a solution combining the dentist's expertise with that of the diabetologist. This would be based on analysis of a photograph of the patient's oral cavity, taken in the department. So far, no studies have ever evaluated the performance of an expert dentist for diagnosing periodontitis from a simple photograph made by non-dental experts in a diabetic department.

The hypothesis is that the concordance in the diagnosis of periodontitis between an indirect method based on a photograph of the oral cavity and a direct method based on clinical examination of this oral cavity (reference) in the diabetic patient would be satisfactory.

DETAILED DESCRIPTION:
Among the complications of diabetes, periodontitis, an infectious disease that destroys the bone and gums, has a bidirectional relationship with diabetes. Indeed, studies have shown that diabetes favors periodontitis, and that periodontitis contributes to the aggravation of diabetes. In addition, the positive impact of treating periodontitis on the indicators and cost of diabetes management has been demonstrated. To echo these findings, since 2020, the French national health scheme now fully covers the treatment of periodontitis in diabetic patients. Unfortunately, health insurance reports point out that 80% of diabetic patients do not visit their dentist enough.

This makes it difficult to detect and treat periodontitis in diabetic patients at an early stage. At the same time, diabetologists who regularly see their patients confirm the importance of knowing their periodontal condition. But they do not have the expertise to diagnose periodontitis whereas, in most cases, a specialist dentist could diagnose it just by looking. The development of a solution allowing the dentist's expertise to be brought to the service of diabetes may have a positive impact on the management of diabetic patients with periodontitis. This expertise could be based on analyzing a photograph of the patient's oral cavity, taken in the department. So far, no studies have ever evaluated the performance of an expert dentist for diagnosing periodontitis from a simple photograph, made by non-dental experts in a diabetic department.

The hypothesis is that the concordance in the diagnosis of periodontitis between an indirect method based on a photograph of the oral cavity and a direct method based on clinical examination of this oral cavity (reference) in the diabetic patient would be satisfactory.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or 2 diabetes.
* Patients of legal age (≥ 18 years).
* Patient undergoing day or weekday hospitalization in the Metabolic and Endocrine Diseases Department at Nîmes University Hospital.
* Patient who has not reported his or her opposition to participating in the study.
* Patient affiliated or beneficiary of a health insurance plan.

Exclusion Criteria:

* Patient who has received treatment for periodontal disease within the past 12 months.
* Patient with fewer (<) than 3 functional contiguous teeth.
* Patient participating in research involving human subjects defined as category 1.
* Patient in an exclusion period as determined by another study.
* Patient under court protection, guardianship, or conservatorship.
* Patient for whom informed information cannot be provided.
* Patient who is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Parodontitis based on a photograph of the patient's oral cavity (indirect method) | Day 0 to day 7
  For the indirect method, two expert dentists will independently analyze the photographs in order to decide whether YES / NO the patient has parodontitis.
Parodontitis based on clinical observation of the patient's oral cavity (direct method) | Day 0
  For the direct method by clinical examination, an expert dentist different from those involved in the indirect method will decide whether YES / NO the patient has parodontitis.

SECONDARY OUTCOMES:
A. Sensitivity and specificity of the Positive Predictive Value (NPV) measured by the indirect method | Day 0 to day 7
  Positive predictive value = True Positive / (True Positives+False Positives)
A. Sensitivity and specificity of the Negative Predictive Value (NPV) measured by the indirect method | Day 0 to day 7
  Negative predictive value = True Negative / (False Negatives + True Negatives)
A. Sensitivity and specificity of the Positive Predictive Value (PPV) measured by the direct method | Day 0
  Positive predictive value = True Positive / (True Positives+False Positives)
A. Sensitivity and specificity of the Positive Predictive Value (PPV) measured by the indirect method | Day 0 to day 7
  Negative predictive value = True Negative / (False Negatives+True Negatives)
B. Quality of photographs taken by the diabetology department : respect of anonymity | Day 0 to day 7
  Evaluation of the photograph by two expert dentists who check compliance with the rules established for taking the photo.
  During the research or at its conclusion, the data collected on the persons who lend themselves to it and transmitted to the sponsor by the investigators (or any other specialized intervening parties) will be made anonymous. Under no circumstances will the names of the persons concerned or their addresses appear in clear text. The patient will be identified only by a unique seven-digit identification number. A list of subject identifications will be kept in the investigator's file. The investigator will ensure that the anonymity of each individual participating in the study is guaranteed. No identifying information will be given to any third party other than those who are authorized by law to hold such information (and who are bound by professional secrecy).
B. Quality of photographs taken by the diabetology department : visibility of the gums | Day 0 to day 7
  Two expert dentists will check compliance with the rules established for taking the photo. For sufficient diagnostic quality, the gums must be clearly visible. "Periodontal disease" describes all gingivitis and periodontitis. Gingivitis is characterized by gingival inflammation manifested by redness of the gums, bleeding and localized edema. The inflammatory process only affects the superficial periodontium (gingival epithelium and gingival connective tissue) and is most often due to an accumulation of bacterial plaque. However, it can be reversed with specific oral hygiene measures. When the deep periodontal tissues (alveolar bone, periodontal ligament, cementum) are affected it is called periodontitis. These lesions are clinically characterized by gingival inflammation and a periodontal pocket (space that is created between the tooth and the gum) as well as by bone loss.
B. Quality of photographs taken by the diabetology department : image sharpness | Day 0 to day 7
  Evaluation of the photograph by two expert dentists who check compliance with the rules established for taking the photo. Is the image sharpness good enough to clearly visualize the patient's gums? YES/NO
B. Quality of photographs taken by the diabetology department : use of the flash | Day 0 to day 7
  Evaluation of the photograph by two expert dentists who check compliance with the rules established for taking the photo. Was the flash used ? YES/NO
B. Quality of photographs taken by the diabetology department : absence of zoom | Day 0 to day 7
  Evaluation of the photograph by two expert dentists who check compliance with the rules established for taking the photo.Was the zoom used? YES/NO
B. Quality of photographs taken by the diabetology department : orientation | Day 0 to day 7
  Evaluation of the photograph by two expert dentists who check compliance with the rules established for taking the photo. Was the photo taken from full front view ? YES/NO
B. Percentage of photographs meeting all of the above criteria for acceptance | Day 0 to day 7
  The number of photographs that meet all the above acceptance criteria will be converted into a percentage.
C. Association between the patient's diabetic constants and his/her periodontal status. Hospitalization | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  - the type of hospitalization (day or week)
C. Association between the patient's diabetic constants and his/her periodontal status. Type of diabetes | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  -the type of diabetes (Type I, Type II or other)
C. Association between the patient's diabetic constants and his/her periodontal status. Age of diabetes | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  - Age of diabetes: <1 year, 1-5 years, 5-10 years, 10-20 years, >20 years
C. Association between the patient's diabetic constants and his/her periodontal status. Treatment | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  -treatment: insulin therapy yes/no and the drug used (metformin, hypoglycemic sulfonamides, dipeptidyl peptidase IV inhibitors, SGLT2 inhibitors, GLP1 analogues, other) will be recorded.
C. Association between the patient's diabetic constants and his/her periodontal status.HbA1c level | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  - the patient's HbA1c level will be recorded in mmol/mol
C. Association between the patient's diabetic constants and his/her periodontal status. Macrovascular complications | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  -Presence of macrovascular complications will be recorded as YES/NO
C. Association between the patient's diabetic constants and his/her periodontal status. Type of macrovascular complication | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  -The type of macrovascular complication : arteriopathy (cerebral, coronary, lower limbs) will be recorded
C. Association between the patient's diabetic constants and his/her periodontal status. Microvascular complications | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  -presence of microvascular complications, YES/NO
C. Association between the patient's diabetic constants and his/her periodontal status. Type of microvascular complication | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  -The type of microvascular complication (retinopathy, nephropathy, neuropathy) will be recorded
C. Association between the patient's diabetic constants and his/her periodontal status. Smoking | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  - the patient's smoking status (active/number of cigarettes per day/ex-smoker) will be recorded
C. Association between the patient's diabetic constants and his/her periodontal status. Periodontitis | Day 0
  Diabetic findings according to the following criteria recorded for each patient included:
  Presence of periodontitis (yes/no) according to the reference method, i.e. by odontological examination.
D. Visible clinical signs associated with periodontitis on the photos taken. Inflammation | Day 0 to day 7
  Evaluation of clinical signs visible on the photos of diabetic patients diagnosed with periodontitis according to the gold standard (odontological examination):
  -Inflammatory color of the gum The evaluation will be interpreted by two blinded expert dentists (different from the one who performed the odontological examination) at the end of the inclusion period.
  Observation of the photographs by two expert dentists.
D. Visible clinical signs associated with periodontitis on the photos taken. Root tartar | Day 0 to day 7
  Evaluation of clinical signs visible on the photos of diabetic patients diagnosed with periodontitis according to the gold standard (odontological examination):
  -Root tartar The evaluation will be interpreted by two blinded expert dentists (different from the one who performed the odontological examination) at the end of the inclusion period.
  Observation of the photographs by two expert dentists.
D. Visible clinical signs associated with periodontitis on the photos taken. Pus | Day 0 to day 7
  Evaluation of clinical signs visible on the photos of diabetic patients diagnosed with periodontitis according to the gold standard (odontological examination):
  -Pus The evaluation will be interpreted by two blinded expert dentists (different from the one who performed the odontological examination) at the end of the inclusion period.
  Observation of the photographs by two expert dentists.
D. Visible clinical signs associated with periodontitis on the photos taken. Bleeding | Day 0 to day 7
  Evaluation of clinical signs visible on the photos of diabetic patients diagnosed with periodontitis according to the gold standard (odontological examination):
  -Bleeding The evaluation will be interpreted by two blinded expert dentists (different from the one who performed the odontological examination) at the end of the inclusion period.
  Observation of the photographs by two expert dentists.
D. Visible clinical signs associated with periodontitis on the photos taken. Interdental space | Day 0 to day 7
  Evaluation of clinical signs visible on the photos of diabetic patients diagnosed with periodontitis according to the gold standard (odontological examination):
  -Interdental space The evaluation will be interpreted by two blinded expert dentists (different from the one who performed the odontological examination) at the end of the inclusion period.
  Observation of the photographs by two expert dentists.
D. Visible clinical signs associated with periodontitis on the photos taken. Gum retraction | Day 0 to day 7
  Evaluation of clinical signs visible on the photos of diabetic patients diagnosed with periodontitis according to the gold standard (odontological examination):
  -Retraction of the gum The evaluation will be interpreted by two blinded expert dentists (different from the one who performed the odontological examination) at the end of the inclusion period.
  Observation of the photographs by two expert dentists.
D. Visible clinical signs associated with periodontitis on the photos taken. Swollen gums | Day 0 to day 7
  Evaluation of clinical signs visible on the photos of diabetic patients diagnosed with periodontitis according to the gold standard (odontological examination):
  -Gum swelling The evaluation will be interpreted by two blinded expert dentists (different from the one who performed the odontological examination) at the end of the inclusion period.
  Observation of the photographs by two expert dentists.
D. Visible clinical signs associated with periodontitis on the photos taken. Plaque | Day 0 to day 7
  Evaluation of clinical signs visible on the photos of diabetic patients diagnosed with periodontitis according to the gold standard (odontological examination):
  -Dental plaque The evaluation will be interpreted by two blinded expert dentists (different from the one who performed the odontological examination) at the end of the inclusion period.
  Observation of the photographs by two expert dentists.

OTHER OUTCOMES:
Sex of patients | Day 0
  Male/female
Age of patients | Day 0
  In years
Type of hospitalization | Day 0
  Inpatients/Outpatients
Periodontal status | Day 0
  Periodontitis / gingivitis / healthy
Lifestyle | Day 0
  Lives alone / Lives with family or nearby / Homeless
Level of education | Day 0
  Primary / Secondary / Graduate / Post-graduate
Professional activity | Day 0
  Employed / Full-time/ Part-time/ Unemployed
Type of diabetes | Day 0
  Type 1 / Type 2 / Unknown / Other
Diabetic for how long | Day 0
  More than 20 years / 10 to 20 years / 5 to 10 years / Less than 5 years / Unknown
Presence of microangiopathic complications | Day 0
  YES / NO
Presence of retinopathy | Day 0
  YES / NO / Don't know
Presence of nephropathy | Day 0
  YES / NO / Don't know
Presence of peripheral neuropathy | Day 0
  YES / NO / Don't know
Glomerular filtration rate (GFR) | Day 0
  GFR between 60 and 89 ml/min/1.73 m² GFR between 45 and 59 ml/min/1.73 m² GFR between 30 and 44 ml/min/1.73 m² GFR between 15 and 29 ml/min/1.73 m² GFR < 15 ml/min/1.73 m²
Dialysis | Day 0
  YES / NO
Presence of macroangiopathic complications | Day 0
  YES / NO
Presence of obliterative arteritis of the lower limbs | Day 0
  YES / NO / Don't know
Presence of supra-aortic arterial trunk disease | Day 0
  YES / NO / Don't know
Presence of coronary artery disease | Day 0
  YES / NO / Don't know
Oral treatment for diabetes | Day 0
  Biguanides / Glucose-lowering sulfonamides / Glinides / Dipeptidyl Peptidase-IV / A-glucosidase inhibitors / SGLT2 inhibitors / None
Injectable antidiabetic treatment | Day 0
  Fast/ultra-fast insulin / Slow/ultra-slow insulin / GLP1 analogues / none
Other treatments | Day 0
  Yes / No If yes specify: Corticosteroids / Chemotherapy / Immunosuppressors / Immunomodulators / Targeted therapy
Weight | Day 0
  In kilos
Height | Day 0
  In centimeters
Body Mass Index | Day 0
  Body Mass Index = kg/m2 where kg is the person's weight in kilograms and m2 is their height in metres squared.
Smoking status | Day 0
  Yes/ No < 10 cigarettes per day
  ≥ 10 cigarettes / day Smoking cessation Yes / No
Alcohol use | Day 0
  Yes / No / Withdrawal
Charlson score | Day 0
  Mild liver disease: Yes / No Moderate to severe liver disease: Yes / No Cerebrovascular disease (excluding hemiplegia): Yes / No Venous insufficiency of the lower limbs: Yes / No Mesenteric vascular disease: Yes / No Renal artery vascular disease: Yes / No Aortic aneurysm : Yes / No Peptic ulcer disease : Yes / No Chronic lung disease : Yes / No Connectivitis: Yes / No Non-metastatic solid tumor : Yes / No Metastatic solid tumor : Yes / No Leukemia : Yes / No Lymphoma, Myeloma: Yes / No AIDS : Yes / No Organ transplant / Yes / No

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nimes, Nîmes, France